CLINICAL TRIAL: NCT05135767
Title: Biobehavioral Pathways Underlying Alcohol Use and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011002840; P20GM130414 (NIH)
Record Dates: First submitted 2021-11-05; First posted 2021-11-26 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Use Disorder; Liver Diseases
Keywords: Alcohol Use Disorder; Liver Diseases; Craving; Ecological Momentary Assessment; Biobehavioral
MeSH Terms: conditions — Alcoholism; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Use Disorder Only (Active Comparator): Individuals in the Alcohol Use Disorder Only arm will meet criteria for alcohol use disorder but will not show evidence of advanced alcohol-associated liver disease. Both arms receive the same brief motivational intervention with personalized feedback.
  Interventions: Behavioral: Brief Motivational Interviewing with Personalized Feedback
- Alcohol Associated Liver Disease + Alcohol Use Disorder (Active Comparator): Individuals in the Alcohol Associated Liver Disease + Alcohol Use Disorder arm will meet criteria for alcohol use disorder and also show evidence of advanced alcohol-associated liver disease. Both arms receive the same brief motivational intervention with personalized feedback.
  Interventions: Behavioral: Brief Motivational Interviewing with Personalized Feedback

INTERVENTIONS:
Behavioral: Brief Motivational Interviewing with Personalized Feedback — A brief motivational interviewing (MI) intervention will target drinking. The intervention will leverage in-depth personalized feedback to identify areas of progress and barriers to change. The personalized feedback will include results of laboratory diagnostic tests, summary reports of timeline followback interviews, and graphical depictions of self-monitoring reports collected on smartphones in daily life. The brief intervention will include an initial 60-minute videoconference session, two brief, 5-10 minute phone-call check-ins completed one and two weeks after the initial intervention, and a 30-minute videoconference booster session completed three weeks after the initial intervention.

SUMMARY:
Alcohol-associated liver disease (ALD) and alcohol use disorder (AUD) are intersecting diseases that add substantially to the global burden of disease and mortality. ALD refers to a spectrum of liver tissue injury caused by chronic and excessive alcohol use. Although reducing drinking is a main treatment goal, this is often unachievable for many patients with ALD due to an underlying AUD characterized by alcohol craving and drinking despite harms. While numerous, high-quality studies demonstrate effectiveness of brief psychosocial interventions for AUD, few trials have tested the efficacy of psychosocial interventions to reduce drinking in individuals with or at risk for ALD. This project establishes a team of addiction scientists and hepatologists to form a partnership and support future collaboration.

DETAILED DESCRIPTION:
The long-term goal of this research program is to develop more effective behavioral interventions to halt the progression of alcohol-associated liver disease (ALD) by addressing at-risk drinking patterns and alcohol use disorder (AUD). The investigators originally proposed a prospective, two-arm intervention study comparing individuals with ALD and AUD vs. those with AUD and without a prior history of ALD or current blood biomarkers suggestive of ALD. The proposed project was designed to demonstrate the feasibility of implementing a brief motivational intervention targeting drinking for patients with ALD recruited from specialty gastroenterology clinics. To keep pace with the original overall recruitment targets within the confines of an adjusted award period, the approach was modified to continue recruiting individuals with AUD and at risk for ALD from the community beyond the original balanced sample size for this group.

After clinic and community recruitment, screening, and enrollment, participants complete four weeks of digital health self-monitoring of precursors of drinking in real-world settings, paired blood biomarkers of liver function, inflammation, and immune response collected prior to the behavioral intervention, at 3 weeks, and at 3-month follow-up. After the first week of self-monitoring, participants attend an in-person research visit involving questionnaires, a laboratory alcohol-cue-reactivity task, and receive a 60-minute, video-conference brief motivational intervention with personalized feedback from self-monitoring reports completed via smartphones in daily life and liver-health biomarkers. The intervention is followed by three weekly research visits culminating with a 30-minute booster video-conference intervention with personalized feedback and exit interviews. A final, in-person research visit is completed at 3 months to evaluate post-intervention, near-term outcomes.

Primarily, this project aims to establish our team and collect initial feasibility and acceptability data for a full-scale clinical trial evaluating biobehavioral endophenotypes AUD in individuals at risk for or with chronic liver disease. At-risk drinking is studied in the setting of a brief intervention designed to enhance knowledge of liver-health risk factors, identify personal precursors of drinking, and increase motivation for sustained change. Secondarily, this project aims to test whether biobehavioral endophenotypes associated with alcohol-use outcomes in clinical trials can serve as indicators of AUD treatment response among individuals at risk for or with ALD. Biomarkers of inflammation and immune activation are explored as mechanisms of persistence of endophenotypes, specifically levels of pro-inflammatory cytokines, chemokines, and others implicated in the pathogenesis of ALD. All study procedures and intervention are offered in English and Spanish, preparing for future full-scale clinical intervention trials among monolingual Spanish-speaking individuals.

ELIGIBILITY:
General Inclusion Criteria. To be eligible, the interested volunteer must:

1. Be at least 18 years of age.
2. Meet the Diagnostic and Statistical Manual-5 criteria for alcohol use disorder, indicated by meeting 2 or more symptom criteria.
3. If male, report 14 or more standard alcoholic drinks per week, or if female, report 7 or more standard alcoholic drinks per week at any point in the 90 days prior to enrollment.
4. Be able to speak and read English or Spanish in order to provide written informed consent and understand written and oral instructions in English or Spanish.

General Exclusion Criteria. Interested volunteers must not have any of the following:

1. Meet the Diagnostic and Statistical Manual-5 criteria for a current diagnosis of psychotic disorders.
2. Currently receiving specialized psychosocial treatment for an alcohol-use or drug problem.
3. If female, pregnant or nursing.
4. Be anyone who, in the opinion of the investigative team, could not currently be safely withdrawn from alcohol without medical detoxification.
5. A BMI of 40 or more, or 35 or more and experiencing obesity-related health conditions, such as high blood pressure or diabetes.
6. Known medical conditions that, in the opinion of the investigative team, would confound results (e.g., uncontrolled infections, multiorgan failure, uncontrolled upper gastrointestinal bleeding, hepatocellular carcinoma or other active malignancies except skin cancer).
7. Patients who have received a liver transplant or are too ill to participate.
8. Pre-existing loss of kidney function with estimated glomerular filtration rate < 30.
9. Any other condition that, in the opinion of the investigative team, would make the interested volunteer unsuitable for the study or unable to comply with the requirements.

Additional Inclusion Criteria for the ALD + AUD Arm.

To be eligible in the ALD+AUD group, the interested volunteer must be diagnosed with advanced alcohol-associated liver disease (i.e., either alcoholic hepatitis or alcoholic cirrhosis). ALD will be determined by chart review. Interested volunteers must have one of the following:

1. Positive liver biopsy, or
2. Fibroscan® score > 12.5, or
3. Evidence of a nodular liver or portal hypertension on abdominal imaging, or
4. Presence of portal hypertensive complications such as hepatic encephalopathy, ascites, or varices, or
5. Fibrosis-4 index >= 3.25, or
6. Aspartate transaminase-platelet ratio index >= 1.0.

Additional Exclusion Criteria for the AUD-only Arm. To be eligible in the AUD-only group, the interested volunteer must not show the following diagnostic test results indicating advanced, alcoholic fibrosis >=F3.

1. Fibrosis-4 index >= 3.25*, or
2. Aspartate transaminase-platelet ratio index >= 1.0**, or
3. Gamma-glutamyl transpeptidase-to-platelet ratio >= 0.32.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Treloar Padovano, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Brown University School of Public Health, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be kept and used for future research on chronic disease and substance use. This includes biospecimens.
Supporting Information: Study Protocol, SAP
Time Frame: Core data including biospecimens collected to fulfill the aims of the Center for Addiction and Disease Risk Exacerbation will be available to request immediately following publication with no prespecified end date. Project-specific data collected to fulfill the research aims outlined in this clinical trial registration will be made available beginning 9 months and ending 36 months following article publication.
Access Criteria: After all data are collected and the results of the study are published, deidentified data and biospecimens may be made available to other qualified investigators at Brown or other institutions upon request. The request will be evaluated by the investigators to ensure that it meets reasonable demands of scientific integrity.

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Alcohol Use Disorder Only | Alcohol Associated Liver Disease + Alcohol Use Disorder
Started | 29 (The "Started" value reflects 29 interested volunteers who were eligible at screening and completed informed consent in the AUD-only group. One was lost to contact prior to completing baseline assessments, and 28 (97%) completed baseline.) | 8 (The "Started" value reflects 8 interested volunteers who were eligible at screening and completed informed consent in the AUD+ALD group. Two withdrew prior to completing baseline assessments, one was lost to contact prior to completing baseline assessments, and 5 (63%) completed baseline.)
Completed | 28 | 5
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Active Study Phase
Arm/Group | Alcohol Use Disorder Only | Alcohol Associated Liver Disease + Alcohol Use Disorder
Started | 28 | 5
Week 1 | 27 | 5
Week 2 | 27 | 5
Completed (Week 3) | 26 | 5
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: The "Overall Number of Baseline Participants" is the count of participants who were included in analyses addressing primary aims. Since Aim 1 evaluates the feasibility of retention between "Screening" and "Baseline" visits, this overall number is the count of participants who were eligible at the "Screening" visit. For ease of interpretation, the participant flow may be viewed as a multiple baseline design, with the "Screening" visit interpreted as "Baseline 1" and "Baseline" as "Baseline 2."
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol Use Disorder Only | Alcohol Associated Liver Disease + Alcohol Use Disorder | Total
Number analyzed (Participants) | 29 | 8 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 4 | 33
  >=65 years | 0 | 4 | 4
Age, Continuous [Mean (Full Range); unit: years] | 44.3 [21 to 63] | 58.3 [33 to 80] | 47.3 [21 to 80]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender, Customized: Cisgender Man | 14 | 7 | 21
  Sex/Gender, Customized: Cisgender Woman | 14 | 1 | 15
  Sex/Gender, Customized: Transgender Woman | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 2 | 11
  Not Hispanic or Latino | 19 | 6 | 25
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 15 | 6 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 9 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 29 | 8 | 37
Recruitment Source [Count of Participants; unit: Participants]
  Community | 29 | 1 | 30
  Clinic | 0 | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Screen Eligible Who Enroll
Description: Feasibility will be evaluated through the percentage of those who are screened as eligible for the study who enroll as participants in the study. The target enrollment rate is greater than or equal to 60% of screen eligible.
Time Frame: 3 months
Population: Overall Number of Participants Analyzed in each Arm/Group is the number of participants who screened eligible for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol Use Disorder Only | Alcohol Associated Liver Disease + Alcohol Use Disorder
Number analyzed (Participants) | 29 | 8
Participants | 28 | 5

2. Primary Outcome: Percentage of Participants Who Complete the Study
Description: Feasibility will be evaluated through the percentage of those participants who are enrolled in the study who complete the study. The target retention rate is greater than or equal to 70% of enrolled participants.
Time Frame: 3 months
Population: Overall Number of Participants Analyzed in each Arm/Group is the number of participants who enrolled in the study, defined as screening eligible and completing baseline assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol Use Disorder Only | Alcohol Associated Liver Disease + Alcohol Use Disorder
Number analyzed (Participants) | 28 | 5
Participants | 26 | 5

3. Primary Outcome: Percentage of Participants Who Withdraw
Description: Acceptability will be evaluated through the percentage of those participants who enroll in the study who withdraw from the study. A participant is considered to have withdrawn from the study if they indicate that they no longer wish to be a part of the study (i.e., not lost to contact). The target withdrawal rate is less than or equal to 20% of enrolled participants.
Time Frame: 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol Use Disorder Only | Alcohol Associated Liver Disease + Alcohol Use Disorder
Number analyzed (Participants) | 28 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 90 days following Baseline assessments.
Arm/Group | Alcohol Use Disorder Only | Alcohol Associated Liver Disease + Alcohol Use Disorder
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/8
Other Adverse Events (participants affected / at risk) | 0/29 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT05135767/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT05135767/SAP_001.pdf
  • Informed Consent Form (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT05135767/ICF_002.pdf